CLINICAL TRIAL: NCT05188144
Title: Early Treatment of Heart Failure: a Non-interventional Observational Study Program of Patients With Heart Failure and Initiated on Dapagliflozin (EVOLUTION-HF - UK)
Brief Title: Real-world Dapagliflozin Experience in Patients With Heart Failure in United Kingdom.
Acronym: EVOLUTION-HF
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D169CR00001
Record Dates: First submitted 2021-11-09; First posted 2022-01-12 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Heart failure (HF) is a global, public health issue that affects more than 63 million people worldwide; this burden is expected to increase substantially as the population ages. Despite advancements in treatment, a HF diagnosis still leads to significant morbidity and mortality; there is also an immense impact on patients' health-related quality of life (HRQoL). On May 5, 2020, the US Food and Drug Administration (FDA) announced the approval of dapagliflozin for heart failure with reduced ejection fraction (HFrEF), regardless of whether the patient has diabetes. Subsequently, there have been additional approvals for this indication by regulatory authorities across the globe." Real-world observational data are necessary to describe dapagliflozin use in real-world settings with detailed clinical data on heart failure symptoms, outcomes, and HRQoL

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years as of study index date; the study index date is date of initiation of treatment with dapagliflozin
* Patient received/receiving treatment with dapagliflozin for HFrEF (EF ≤40%) in accordance with the local dapagliflozin product label
* Signed and dated informed consent prior to enrolment in the study

Exclusion Criteria:

* Patient is enrolled less than 14 days or more than 60 days following initiation of dapagliflozin
* Prior treatment with dapagliflozin or other SGLT2i treatment
* Initiation of dapagliflozin outside of local HF label
* Diagnosis of Type 1 diabetes prior to enrolment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have received treatment with dapagliflozin for HFrEF will be eligible for enrolment by either primary or secondary care healthcare professionals from both outpatient and inpatient settings. In all cases, the decision to treat a patient with dapagliflozin must be made prior to the decision to enrol the patient into the study. To help ensure this, patients cannot be enrolled <14 days after starting dapagliflozin treatment. Therefore, the earliest date at which all data collected directly from patients such as PROs may be captured is 14 days following initiation of dapagliflozin. Patients may have discontinued from dapagliflozin prior to enrolment onto the study, as long as their dapagliflozin initiation was ≥14 days and ≤60 days prior to enrolment onto the study. Data on other parameters may be obtained at the date of initiation of dapagliflozin by extracting this information retrospectively from medical charts.
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2024-03-02 (Actual); Study Completion 2024-03-02 (Actual)

PRIMARY OUTCOMES:
Time to dapagliflozin treatment discontinuation | Baseline to 12 months
  Time from dapagliflozin treatment initiation until the time at which participants stop taking the medication for any reason.
Number of reasons for dapagliflozin treatment discontinuation | Baseline to 12 months
  Number of reason for dapagliflozin treatment discontinuation as noted by a health care professional will extracted and described as the number and proportion of participants who have discontinued dapagliflozin according to each reasons presented.
Proportion of reasons for dapagliflozin treatment discontinuation | Baseline to 12 months
  Proportion of reasons for dapagliflozin treatment discontinuation as noted by a health care professional will extracted and described as the number and proportion of participants who have discontinued dapagliflozin according to each reasons presented.
Number of dapagliflozin treatment changes | Baseline to 12 months
  The number of participants who switch to another HF medication other than dapagliflozin.
Percentage of dapagliflozin treatment changes | Baseline to 12 months
  The percentage of participants who switch to another HF medication other than dapagliflozin.
Number of dapagliflozin treatment discontinuation | Baseline to 12 months
  The number of participants who discontinued treatment with dapagliflozin.
Percentage of dapagliflozin treatment discontinuation | Baseline to 12 months
  The percentage of participants who discontinued treatment with dapagliflozin.
Time to other heart failure treatment discontinuation | Baseline to 12 months
  Time from initiation of heart failure medication other than dapagliflozin until the time at which participants discontinued treatment with that medication.
Number of other heart failure treatment initiation | Baseline to 12 months
  The number of participants who initiate new heart failure medication other than dapagliflozin.
Percentage of other heart failure treatment initiation | Baseline to 12 months
  The percentage of participants who initiate new heart failure medication other than dapagliflozin.
Number of other heart failure treatment dosage changes | Baseline to 12 months
  The number of participants with dosage changes for heart failure medication other than dapagliflozin.
Percentage of other heart failure treatment dosage changes | Baseline to 12 months
  The percentage of participants with dosage changes for heart failure medication other than dapagliflozin.
Number of other heart failure treatment discontinuation | Baseline to 12 months
  The number of participants who discontinue treatment with heart failure medication other than dapagliflozin.
Percentage of other heart failure treatment discontinuation | Baseline to 12 months
  The percentage of participants who discontinue treatment with heart failure medication other than dapagliflozin.
Time to glucose lowering medication discontinuation | Baseline to 12 months
  Time from initiation of glucose lowering medication other than dapagliflozin until the time at which participants discontinued treatment with that medication.
Number of glucose lowering medication initiation | Baseline to 12 months
  The number of participants who initiate new glucose lowering medication other than dapagliflozin.
Percentage of glucose lowering medication initiation | Baseline to 12 months
  The percentage of participants who initiate new glucose lowering medication other than dapagliflozin.
Number of glucose lowering medication dosage changes | Baseline to 12 months
  The number of participants with dosage changes for glucose lowering medication other than dapagliflozin.
Percentage of glucose lowering medication dosage changes | Baseline to 12 months
  The percentage of participants with dosage changes for glucose lowering medication other than dapagliflozin.
Number of glucose lowering medication discontinuation | Baseline to 12 months
  The number of participants who discontinue treatment with glucose lowering medication other than dapagliflozin.
Percentage of glucose lowering medication discontinuation | Baseline to 12 months
  The percentage of participants who discontinue treatment with glucose lowering medication other than dapagliflozin.

SECONDARY OUTCOMES:
Absolute change from baseline in Kansas City Cardiomyopathy Questionnaire (KCCQ) score | Measured at 3, 6, 9 and 12 months
  The KCCQ is a 23-item questionnaire that quantifies physical limitations, self-efficacy, social interference and quality of life. Summary scores will be examined at each assessment point during follow-up. For each of the assessment periods, descriptive statistics for the observed value, change from baseline and the 95% two-sided confidence interval for the mean change will be presented. The proportions of participants with overall health status classified as poor, fair, good, and excellent will be examined at each assessment point. Additionally, the proportions of participants who experience clinically meaningful changes in overall health status: improvement (≥5 point increase), deterioration (≥5 point decrease), and stable (<5 point increase or decrease) will be examined at each assessment point.
Absolute change from baseline in Medication Adherence Report Scale (MARS)-5 questionnaire | Measured at 3, 6, 9 and 12 months
  The MARS-5 is five-item self-report adherence scale which assesses both intentional and non-intentional non-adherence. Respondents rate the frequency with which the five different medication-taking behaviours occur, scoring each item on a 1-5-point scale with higher scores indicating higher reported adherence. The MARS-5 has been shown to be reliable and valid across a variety of health conditions, including cardiovascular and pulmonary diseases.
Absolute change from baseline in Work Productivity and Activity Impairment (WPAI) score | Measured at 3, 6, 9 and 12 months
  The WPAI is a validated instrument to measure impairments in paid and unpaid work and activities. It measures absenteeism (work time missed), presenteeism (impairment at work / reduced on-the-job effectiveness) as well as the impairments in unpaid activity because of health problems during the past seven days. It has been validated to quantify work impairments for numerous diseases such as asthma, psoriasis, irritable bowel syndrome, and Crohn's disease, but has not yet been validated for use in heart failure participants. Scores will be derived from the overall work impairment at each timepoint and then changes of from baseline will be reported.

CONTACTS AND LOCATIONS:
Locations (10):
- United Kingdom (10):
  - Research Site, Reading, Berkshire
  - Research Site, Truro, Cornwall
  - Research Site, Portadown, County Armagh
  - Research Site, Barnstaple, Devon
  - Research Site, Westcliff-on-Sea, Essex
  - Research Site, Port Talbot, Glamorgan
  - Research Site, London, Greater London
  - Research Site, Stoke-on-Trent, Staffordshire
  - Research Site, Brighton, Sussex
  - Research Site, Coventry, Warwickshire

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D169CR00001&attachmentIdentifier=2ebb8e94-a77a-42d3-9465-470af0b756ea&fileName=D169CR00001_Redacted_CSR_Synopsis.pdf&versionIdentifier=